CLINICAL TRIAL: NCT01950598
Title: Boston Keratoprosthesis Type 1 Surgery: Use of Frozen Versus Fresh Corneal Donor Carriers
Brief Title: Frozen Versus Fresh Corneal Carriers for the Boston KPro Type I Donor Carriers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie-Claude Robert (Other)
Collaborators: Fonds de recherche en ophtalmologie de l'Université de Montréal (Other)
Responsible Party: Sponsor-Investigator, Marie-Claude Robert, MD, FRSCS, Centre hospitalier de l'Université de Montréal (CHUM)
Organization: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FvF 08.275
Record Dates: First submitted 2013-09-09; First posted 2013-09-25 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Corneal Blindness; Boston Keratoprosthesis Type I Candidate
Keywords: Boston Keratoprosthesis type I surgery, frozen corneal graft

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fresh carrier graft for KPro (Active Comparator): KPro implanted using fresh cornea, preserved in optisol GS
  Interventions: Procedure: Boston KPro type I - fresh graft
- Frozen carrier graft for KPro (Experimental): KPro implanted using frozen cornea, which was supplied as a whole globe cryopreserved at -80°C in gramicidin 0.025 mg/mL and polymyxin B sulfate 10 000 U/mL ophthalmic solution.
  Interventions: Procedure: Boston KPro type I surgery - frozen graft

INTERVENTIONS:
Procedure: Boston KPro type I - fresh graft — Boston KPro mounted on fresh corneal carrier graft for implantation
  Arms: Fresh carrier graft for KPro
Procedure: Boston KPro type I surgery - frozen graft — Boston KPro mounted on frozen corneal carrier graft for implantation
  Arms: Frozen carrier graft for KPro

SUMMARY:
The purpose of this study is to determine whether frozen corneas are as safe and effective as fresh corneas for use as carriers with the Boston Keratoprosthesis type I (KPro) over long term follow-up.

Corneal transplantation is typically performed using fresh, transparent corneas. With KPro surgery, the corneal transplant only serves as a carrier to suture the KPro in place. The cornea used in KPro surgery does not need to be clear like a normal transplant. Frozen corneal tissue can be used to repair the cornea in cases of emergency but the tissue is not transparent and does not allow good vision. We hypothesize that frozen grafts are equivalent as fresh grafts when used as carrier for the KPro.

DETAILED DESCRIPTION:
The Boston Keratoprosthesis (KPro) is a collar-button shaped device made from a specialized clear plastic material. This device is used to replace a diseased and opaque cornea with a clear window so that vision can be improved. KPro surgery is an alternative to a traditional corneal graft and is used when a traditional corneal graft has failed or has a very poor probability of success.

During KPro surgery, the KPro needs to be incorporated into a corneal graft before it is sutured to the patient's cornea. The corneal graft serves as a support to the KPro and helps to re-establish vision. The corneas typically used as carriers for the KPro are fresh corneas provided through donors. These fresh corneas are also used in traditional corneal transplantation, without KPro implantation.

Due to shortage of fresh corneas in the province of Quebec, this project is interested in evaluating if corneas that have been previously frozen can act as carriers to the KPro. The frozen corneas cannot be used in traditional corneal transplantation surgery because they are not transparent. However, they can act as a support to the KPro, as in this case, it is the KPro and not the corneal graft that re-establishes vision. The use of frozen corneas for KPro surgery has the potential to improve access to corneal donor tissue and improve the wait-times for KPro surgery.

37 patients were be recruited from the Centre Hospitalier de l'Université de Montréal (CHUM), Notre-Dame Hospital between October 2008 and November 2009. Participants were divided into 2 groups: the first group will receive a KPro in a fresh corneal carrier graft while the second group will receive a KPro in a frozen carrier graft. The use of a fresh or frozen corneal graft depended on the availability of fresh tissue on the morning of surgery. 19 patients received a fresh carrier graft and 18 received a frozen carrier graft.

Patients were followed on postoperative day 1, week 1 and 2, month 1, 3 and 6 and every 1 to 3 months thereafter up to 2 years. At each follow-up visit, a complete ophthalmological examination was performed, including best-corrected Snellen visual acuity and slit lamp assessment for leaks, tissue necrosis, melts, extrusion, inflammation, retroprosthetic membrane formation and infectious endophthalmitis.

The current study aims re-consent patients previously enrolled in this study to prospectively evaluate the long-term outcomes of KPro surgery using either a fresh or frozen carrier graft. IRB approval was obtained from the CHUM. Written informed consent from the concerned patients will be obtained for this extension study during their routine visits at the CHUM Ophthalmology department.

Patients in this study will continue their routine follow-up at the frequency determined by their surgeon, which may vary from every 3 to 6 months.

Outcome measures include surgical feasibility, level of preoperative and postoperative visual acuity (VA), retention of the device and complications as stated above. Outcomes will be compared at 5 and 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject over age 18 years
* Boston KPro type I indicated
* history, slit-lamp findings and B-scan do not suggest endstage glaucoma or significant posterior segment disease
* Able to provide informed consent for study inclusion
* Sufficiently healthy to undergo surgery and a vigorous post-operative follow-up course
* Able to administer eye medications or have a care-giver able and willing to do the same
* Corneal blindness with poor prognosis for survival of a traditional penetrating keratoplasty

Exclusion Criteria:

* Subject under age 18 years
* History, slit-lamp findings and B-scan suggest endstage glaucoma or significant posterior segment disease
* Not sufficiently healthy to undergo surgery and a vigorous post-operative follow-up course
* Unable to administer eye medication or does not have a care-giver willing to do the same

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Extrusion rate | 10 years post-KPro implantation

SECONDARY OUTCOMES:
Best-corrected visual acuity | 10 years
Retroprosthetic membrane formation | 10 years
Endophthalmitis rate | 10 years
Sterile vitritis rate | 10 years
Intraoperative complications | time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mona Harissi-Dagher, M.D., Principal Investigator — CHUM - Hôpital Notre-Dame
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Result] Robert MC, Biernacki K, Harissi-Dagher M. Boston keratoprosthesis type 1 surgery: use of frozen versus fresh corneal donor carriers. Cornea. 2012 Apr;31(4):339-45. doi: 10.1097/ICO.0b013e31823e6110. PMID 22269678